CLINICAL TRIAL: NCT02310906
Title: A 2-Part, Randomized, Double-Blind, Placebo-Controlled, Dose-Titration, Safety, Tolerability, and Pharmacokinetics Study (Part 1) Followed by an Open-Label Efficacy and Safety Evaluation (Part 2) of SRP-4053 in Patients With Duchenne Muscular Dystrophy Amenable to Exon 53 Skipping
Brief Title: Phase I/II Study of SRP-4053 in DMD Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Collaborators: Institut de Myologie, France (Other); Consultants for Research in Imaging and Spectroscopy (Other); Great Ormond Street Hospital for Children NHS Foundation Trust (Other); Catholic University of the Sacred Heart (Other); Royal Holloway University (Other); SYSNAV (Industry); University College, London (Other); University of Newcastle Upon-Tyne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4053-101
Record Dates: First submitted 2014-12-03; First posted 2014-12-08 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne muscular dystrophy; Exon Skipping; DMD; Exon 53; Ambulatory; Pediatric
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking Description: Part 1 is double-blind and randomized; Part 2 is open-label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: SRP-4053 (Experimental): Patients will receive SRP-4053 (golodirsen) intravenous (IV) infusions, weekly, at escalating dose levels as follows: Weeks 1-2, 4 mg/kg/week; Weeks 3-4, 10 mg/kg/week; Weeks 5-6, 20 mg/kg/week; Weeks 7-12, 30 mg/kg/week. Dosing will be interrupted or halted if specific predefined stopping criteria are met or if warranted at the discretion of the Sponsor or Investigator.
  Interventions: Drug: SRP-4053
- Part 1: Placebo (Placebo Comparator): Patients will receive SRP-4053 placebo-matching IV infusions, weekly, for 12 weeks. Dosing will be interrupted or halted if specific predefined stopping criteria are met or if warranted at the discretion of the Sponsor or Investigator.
  Interventions: Drug: Placebo
- Part 2: SRP-4053 (Experimental): All eligible patients from Part 1, as well as new patients, will receive SRP-4053 (golodirsen) 30 mg/kg/week IV infusions, weekly, for up to 168 weeks.
  Interventions: Drug: SRP-4053
- Part 2: Untreated Group (No Intervention): Patients with DMD who have a genotypically confirmed deletion of exon(s) not amenable to treatment by exon 53 skipping, but who otherwise meet the same eligibility criteria as treated patients newly recruited to Part 2, will undergo the same study assessments as treated Patients (except for pharmacokinetic [PK] sampling and muscle biopsies), but at a reduced schedule through Week 144. The untreated patients are not considered as control group.

INTERVENTIONS:
Drug: Placebo — SRP-4053 placebo-matching solution for IV infusion.
  Arms: Part 1: Placebo
Drug: SRP-4053 — SRP-4053 (golodirsen) solution for IV infusion.
  Arms: Part 1: SRP-4053; Part 2: SRP-4053

SUMMARY:
This is a first-in-human, multiple-dose 2-part study to assess the safety, tolerability, efficacy, and pharmacokinetics of SRP-4053 in Duchenne muscular dystrophy (DMD) patients with deletions amenable to exon 53 skipping.

DETAILED DESCRIPTION:
Part 1: Randomized, placebo-controlled dose-titration to assess safety, tolerability and pharmacokinetics of 4 dose levels of SRP-4053 in genotypically-confirmed DMD patients with deletions amenable to exon 53 skipping.

Part 2: Open-label evaluation of SRP-4053 in patients from Part 1, along with newly enrolled DMD patients with deletions amenable to exon 53 skipping and an untreated group of DMD patients with deletions not amenable to exon 53 skipping.

Safety, including adverse event monitoring and routine laboratory assessments, will be followed on an ongoing basis for all patients.

Clinical efficacy, including functional tests such as the six-minute walk test (6MWT), will be assessed at regularly scheduled study visits. Patients in the treated groups will undergo one baseline and one follow-up muscle biopsy. Patients in the untreated group will not undergo biopsies and will follow an abbreviated schedule of study assessments.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with DMD, genotypically confirmed.
* Intact right and left biceps muscles or an alternative upper arm muscle group.
* Stable pulmonary and cardiac function.
* Minimum performance on 6MWT, North Star Ambulatory Assessment, and rise (Gowers) test as specified in the study protocol.
* On a stable dose of corticosteroids for at least 6 months.

Exclusion Criteria:

* Previous treatment with the experimental agents BMN-195 (SMT C1100) or PRO053.
* Current or previous treatment with any other experimental treatments within 12 weeks prior to study entry.
* Major surgery within the last 3 months.
* Presence of other clinically significant illness.
* Major change in physical therapy regime within the last 3 months.

Other inclusion and exclusion criteria may apply.

Ages: 6 Years to 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2015-01-13 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sarepta Therapeutics, Inc.
Locations (5):
- Boston Children's Hospital, Boston, Massachusetts, United States
- Institute de Myologie, Paris, France
- Policlinico Universitario A Gemelli, Rome, Italy
- United Kingdom (2):
  - Great Ormond Street Hospital for Children NHS Foundation Trust, London
  - Newcastle University Hospital, Newcastle

REFERENCES:
- [Background] Frank DE, Schnell FJ, Akana C, El-Husayni SH, Desjardins CA, Morgan J, Charleston JS, Sardone V, Domingos J, Dickson G, Straub V, Guglieri M, Mercuri E, Servais L, Muntoni F; SKIP-NMD Study Group. Increased dystrophin production with golodirsen in patients with Duchenne muscular dystrophy. Neurology. 2020 May 26;94(21):e2270-e2282. doi: 10.1212/WNL.0000000000009233. Epub 2020 Mar 5. PMID 32139505
- [Derived] Servais L, Mercuri E, Straub V, Guglieri M, Seferian AM, Scoto M, Leone D, Koenig E, Khan N, Dugar A, Wang X, Han B, Wang D, Muntoni F; SKIP-NMD Study Group. Long-Term Safety and Efficacy Data of Golodirsen in Ambulatory Patients with Duchenne Muscular Dystrophy Amenable to Exon 53 Skipping: A First-in-human, Multicenter, Two-Part, Open-Label, Phase 1/2 Trial. Nucleic Acid Ther. 2022 Feb;32(1):29-39. doi: 10.1089/nat.2021.0043. Epub 2021 Nov 17. PMID 34788571

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 5 sites in the France, Italy, United Kingdom and United States from 13 January 2015 to 25 March 2019.
Pre-assignment Details: Study conducted in 2 parts: Part 1 and Part 2. When Part 1 was completed and cumulative safety data was reviewed by an independent Data Safety Monitoring Board (DSMB), Part 2 was conducted.
Groups:
- Part 1: Placebo: Participants received placebo-matched to golodirsen intravenous (IV) infusions, once weekly up to 12 weeks in Part 1.
- Part 1: Golodirsen: Participants received golodirsen IV infusions, at four dose levels of 4 milligrams per kilograms (mg/kg) once weekly for 2 weeks, followed by 10 mg/kg once weekly for the next 2 weeks (i.e., up to Week 4), followed by 20 mg/kg once weekly for the next 2 weeks (i.e., up to Week 6), followed by 30 mg/kg once weekly from Week 7 to Week 12 in Part 1.
- Part 2a: Total Golodirsen Group: All participants from Part 1 (who previously received placebo or golodirsen) and including additional new participants received golodirsen 30 milligram (mg)/kilogram (kg) once weekly, for up to 168 weeks. Dosing was interrupted or halted when any specific predefined stopping criteria was met or if warranted at the discretion of the Sponsor or Investigator.
- Part 2b: Untreated Group (Natural History of Non-exon 53): Untreated participants intended to evaluate the natural history of the disease with DMD and various genetic mutations (not amenable to exon 53 skipping) were included in this group and did not received any treatment. Participants underwent the same study assessments as treated participants in other reporting groups (except for pharmacokinetic [PK] sampling and muscle biopsies), but at a reduced schedule through Week 144. Thus, the untreated participants were not considered as control group.
Period: Part 1: Double Blind Phase (12 Weeks)
Arm/Group | Part 1: Placebo | Part 1: Golodirsen | Part 2a: Total Golodirsen Group | Part 2b: Untreated Group (Natural History of Non-exon 53)
Started | 4 | 8 | 0 | 0
Received 4 mg/kg | 0 | 8 | 0 | 0
Received 10 mg/kg | 0 | 8 | 0 | 0
Received 20 mg/kg | 0 | 8 | 0 | 0
Received 30 mg/kg | 0 | 8 | 0 | 0
Completed | 4 | 8 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part 2: Open Label Phase (168 Weeks)
Arm/Group | Part 1: Placebo | Part 1: Golodirsen | Part 2a: Total Golodirsen Group | Part 2b: Untreated Group (Natural History of Non-exon 53)
Started | 0 | 0 | 25 (4 participants from Part 1(Placebo) + 8 participants from Part 1(Golodirsen) +13 new participants) | 14
Completed | 0 | 0 | 23 | 6
Not Completed | 0 | 0 | 2 | 8
Not completed — Enrollment in other therapeutic study | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 4
Not completed — Personal reasons | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety set included all randomized participants from Part 1 and all Part 2 participants amenable to exon 53 skipping who received any amount of study drug, and all untreated participants who entered Part 2.
Groups:
- Part 2b: Untreated Group (Natural History of Non-exon 53): Untreated participants intended to evaluate the natural history of the disease with DMD and various genetic mutations (not amenable to exon 53 skipping) were included in this group and did not received any treatment. Participants underwent the same study assessments as treated participants in other reporting groups (except for PK sampling and muscle biopsies), but at a reduced schedule through Week 144. Thus, the untreated participants were not considered as control group.
- Total: Total of all reporting groups
Arm/Group | Part 1: Placebo | Part 1: Golodirsen | Part 2a: Total Golodirsen Group | Part 2b: Untreated Group (Natural History of Non-exon 53) | Total
Number analyzed (Participants) | 4 | 8 | 25 | 14 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: All participants who were previously randomized in Part 1 were moved to Part 2a (after completion of Part 1, n=12) along with 13 new participants. Hence, total number of participants in Part 2a were 25. In Part 2b, 14 untreated new participants were enrolled.
  years
    Part 1: number analyzed (Participants) | 4 | 8 | 0 | 0 | 12
    Part 1 | 7.0 (0.82) | 8.6 (2.07) |  |  | 8.1 (1.88)
    Part 2: number analyzed (Participants) | 0 | 0 | 25 | 14 | 39
    Part 2 |  |  | 8.4 (2.18) | 8.5 (1.91) | 8.4 (2.06)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All participants who were previously randomized in Part 1 were moved to Part 2a (after completion of Part 1, n=12) along with 13 new participants. Hence, total number of participants in Part 2a were 25. In Part 2b, 14 untreated new participants were enrolled.
  Participants
    Part 1: number analyzed (Participants) | 4 | 8 | 0 | 0 | 12
    Part 1: Female | 0 | 0 |  |  | 0
    Part 1: Male | 4 | 8 |  |  | 12
    Part 2: number analyzed (Participants) | 0 | 0 | 25 | 14 | 39
    Part 2: Female |  |  | 0 | 0 | 0
    Part 2: Male |  |  | 25 | 14 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: All participants who were previously randomized in Part 1 were moved to Part 2a (after completion of Part 1, n=12) along with 13 new participants. Hence, total number of participants in Part 2a were 25. In Part 2b, 14 untreated new participants were enrolled.
  Participants
    Part 1: number analyzed (Participants) | 4 | 8 | 0 | 0 | 12
    Part 1: Hispanic or Latino | 1 | 1 |  |  | 2
    Part 1: Not Hispanic or Latino | 1 | 4 |  |  | 5
    Part 1: Unknown or Not Reported | 2 | 3 |  |  | 5
    Part 2: number analyzed (Participants) | 0 | 0 | 25 | 14 | 39
    Part 2: Hispanic or Latino |  |  | 4 | 0 | 4
    Part 2: Not Hispanic or Latino |  |  | 9 | 9 | 18
    Part 2: Unknown or Not Reported |  |  | 12 | 5 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: All participants who were previously randomized in Part 1 were moved to Part 2a (after completion of Part 1, n=12) along with 13 new participants. Hence, total number of participants in Part 2a were 25. In Part 2b, 14 untreated new participants were enrolled.
  Participants
    Part 1: number analyzed (Participants) | 4 | 8 | 0 | 0 | 12
    Part 1: American Indian or Alaska Native | 0 | 0 |  |  | 0
    Part 1: Asian | 0 | 0 |  |  | 0
    Part 1: Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  | 0
    Part 1: Black or African American | 0 | 0 |  |  | 0
    Part 1: White | 3 | 8 |  |  | 11
    Part 1: More than one race | 1 | 0 |  |  | 1
    Part 1: Unknown or Not Reported | 0 | 0 |  |  | 0
    Part 2: number analyzed (Participants) | 0 | 0 | 25 | 14 | 39
    Part 2: American Indian or Alaska Native |  |  | 0 | 0 | 0
    Part 2: Asian |  |  | 0 | 1 | 1
    Part 2: Native Hawaiian or Other Pacific Islander |  |  | 0 | 0 | 0
    Part 2: Black or African American |  |  | 0 | 0 | 0
    Part 2: White |  |  | 23 | 11 | 34
    Part 2: More than one race |  |  | 2 | 2 | 4
    Part 2: Unknown or Not Reported |  |  | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs and TEAEs Leading to Discontinuation
Description: Adverse event (AE) was any untoward medical occurrence in a clinical trial participant, which does not necessarily have a causal relationship with the investigational drug. A Serious adverse event (SAE) was an AE resulting in any of the following outcomes: death; Life-threatening event; Required or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly. TEAEs were defined as AEs that were reported or worsened on or after the start of study drug dosing through 12 weeks. TEAEs included both Serious TEAEs and non-serious TEAEs.
Time Frame: Baseline up to Week 12
Population: Part 1 safety set included all randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Placebo: Participants received placebo-matched to golodirsen IV infusions, once weekly for up to 12 weeks in Part 1.
- Part 1: Golodirsen (4 mg/kg): Participants received golodirsen IV infusions, at dose levels of 4 mg/kg, once weekly for 2 weeks in Part 1.
- Part 1: Golodirsen (10 mg/kg): Participants received golodirsen IV infusions, at a dose levels of 10 mg/kg, once weekly for the next 2 weeks (i.e., up to Week 4) in Part 1.
- Part 1: Golodirsen (20 mg/kg): Participants received golodirsen IV infusions, at a dose level of 20 mg/kg, once weekly for the next 2 weeks (i.e., up to Week 6) in Part 1.
- Part 1: Golodirsen (30 mg/kg): Participants received golodirsen IV infusions, at a dose level of 30 mg/kg, once weekly from Week 7 to Week 12 in Part 1.
Arm/Group | Part 1: Placebo | Part 1: Golodirsen (4 mg/kg) | Part 1: Golodirsen (10 mg/kg) | Part 1: Golodirsen (20 mg/kg) | Part 1: Golodirsen (30 mg/kg)
Number analyzed (Participants) | 4 | 8 | 8 | 8 | 8
Participants
  Participants with TEAE | 4 | 5 | 5 | 3 | 6
  Participants with Serious TEAE | 0 | 0 | 0 | 0 | 0
  Participants with TEAEs leading to discontinuation | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Part 1: Number of Participants With Potentially Clinically Significant (PCS) Laboratory Abnormalities Reported as TEAEs
Description: Laboratory parameters included hematology, serum chemistry (SC), urinalysis and coagulation. Number of participants with at least one potentially clinically significant abnormal finding were reported as TEAEs. The Investigator determined whether abnormal assessment results were potentially clinically significant or not. Potentially clinical significance was defined as any variation in assessment results that had medical relevance resulting in an alteration in medical care.
Time Frame: Baseline up to Week 12
Population: Part 1 safety set included all randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: Golodirsen (4 mg/kg) | Part 1: Golodirsen (10 mg/kg) | Part 1: Golodirsen (20 mg/kg) | Part 1: Golodirsen (30 mg/kg)
Number analyzed (Participants) | 4 | 8 | 8 | 8 | 8
Participants
  Hepatic Chemistry | 0 | 0 | 0 | 0 | 0
  Renal Chemistry | 0 | 0 | 0 | 0 | 0
  Hematology | 2 | 0 | 1 | 0 | 0
  Coagulation | 0 | 0 | 0 | 0 | 0
  Urinalysis | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Part 1: Number of Participants With Potentially Clinically Significant Abnormalities in Vital Signs Reported as TEAEs
Description: Vital sign parameters included systolic blood pressure (SBP), diastolic blood pressure (DBP), heart rate (HR), and body temperature. Number of participants with at least one potentially clinically significant abnormal vital signs findings were reported as TEAEs. The Investigator determined whether abnormal assessment results were potentially clinically significant or not. Potential clinical significance was defined as any variation in assessment results that had medical relevance resulting in an alteration in medical care.
Time Frame: Baseline up to Week 12
Population: Part 1 safety set included all randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: Golodirsen (4 mg/kg) | Part 1: Golodirsen (10 mg/kg) | Part 1: Golodirsen (20 mg/kg) | Part 1: Golodirsen (30 mg/kg)
Number analyzed (Participants) | 4 | 8 | 8 | 8 | 8
Participants | 1 | 3 | 1 | 1 | 4

4. Primary Outcome: Part 1: Number of Participants With Potentially Clinically Significant Abnormalities in Physical Examinations
Description: Physical examinations were performed by the Investigator, or qualified study staff. A full physical examination included a review of general appearance, head, eyes, ears, nose and throat, heart, lungs, abdomen, extremities, skin, lymph nodes, musculoskeletal, and neurological systems. Number of participants with potentially clinically significant abnormalities in physical examinations were reported. Potentially clinically significant abnormalities in physical examinations were based on Investigator's discretion.
Time Frame: Baseline up to Week 12
Population: Part 1 safety set included all randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: Golodirsen (4 mg/kg) | Part 1: Golodirsen (10 mg/kg) | Part 1: Golodirsen (20 mg/kg) | Part 1: Golodirsen (30 mg/kg)
Number analyzed (Participants) | 4 | 8 | 8 | 8 | 8
Participants | 0 | 0 | 2 | 0 | 3

5. Primary Outcome: Part 1: Number of Participants With Potentially Clinically Significant Abnormalities in Electrocardiogram (ECG) Reported as TEAEs
Description: Twelve-lead ECGs were performed at a consistent time of day throughout the study. Electrocardiograms were performed only after the participant was in the supine position, resting, and quiet for a minimum of 15 minutes. The ECG was manually reviewed and interpreted by medically qualified personnel. Number of participants with potentially clinically significant abnormalities in ECG reported as TEAEs presented here. The Investigator determined whether abnormal assessment results were potentially clinically significant or not.
Time Frame: Baseline up to Week 12
Population: Part 1 safety set included all randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: Golodirsen (4 mg/kg) | Part 1: Golodirsen (10 mg/kg) | Part 1: Golodirsen (20 mg/kg) | Part 1: Golodirsen (30 mg/kg)
Number analyzed (Participants) | 4 | 8 | 8 | 8 | 8
Participants | 0 | 1 | 0 | 0 | 0

6. Primary Outcome: Part 1: Number of Participants With Potentially Clinically Significant Abnormalities in Echocardiograms (ECHO)
Description: Standard, 2-dimensional ECHOs were performed at a consistent time of day throughout the study. Cardiac function events included cardiomegaly, tachycardia, and dyspnoea. The ECHO was reviewed and interpreted by medically qualified personnel. Number of participants with potentially clinically significant abnormalities in ECHO were reported.
Time Frame: Baseline up to Week 12
Population: Part 1 safety set included all randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: Golodirsen (4 mg/kg) | Part 1: Golodirsen (10 mg/kg) | Part 1: Golodirsen (20 mg/kg) | Part 1: Golodirsen (30 mg/kg)
Number analyzed (Participants) | 4 | 8 | 8 | 8 | 8
Participants | 0 | 0 | 0 | 0 | 3

7. Primary Outcome: Part 2a: Change From Baseline in the Total Distance Walked During 6-Minute Walk Test (6MWT) at Week 144 in Total Golodirsen Group
Description: 6MWT was performed by standardized procedures for all participants. Participants were asked to walk a set course of 25 meters for 6 minutes (timed), and the distance walked (in meters) was recorded. Change from baseline in 6MWT distance at Week 144 in total golodirsen group was reported.
Time Frame: Baseline and Week 144
Population: Efficacy set consisted of all randomized participants who had at least one post baseline functional assessment. Here, overall number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: meters
Groups:
- Part 2a: Total Golodirsen Group: All participants from Part 1 (who previously received placebo or golodirsen) and including additional new participants received golodirsen 30 mg/kg once weekly, for up to 168 weeks in Part 2. Dosing was interrupted or halted when any specific predefined stopping criteria was met or if warranted at the discretion of the Sponsor or Investigator.
Arm/Group | Part 2a: Total Golodirsen Group
Number analyzed (Participants) | 22
meters | -99.0 (123.75)

8. Primary Outcome: Part 2b: Change From Baseline in the Total Distance Walked During 6-Minute Walk Test (6MWT) at Week 144 in Untreated Group (Non-exon 53 Amenable Participants)
Description: 6MWT was performed by standardized procedures for all participants. Participants were asked to walk a set course of 25 meters for 6 minutes (timed), and the distance walked (in meters) was recorded. Change from baseline in 6MWT distance at Week 144 in untreated group (non-exon 53 amenable participants) was calculated.
Time Frame: Baseline and Week 144
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Part 2b: Untreated Group (Natural History of Non-exon 53)
Number analyzed (Participants) | 6
Meters | -160.8 (162.41)

9. Primary Outcome: Part 2a: Change From Baseline in Dystrophin Protein Levels Determined by Western Blot at Week 48 in Total Golodirsen Group
Description: Change from baseline in dystrophin protein levels (in muscle biopsy samples) was determined by Western blot in total golodirsen group.
Time Frame: Baseline, Week 48
Population: Muscle biopsy set included all participants who received at least one dose of study drug and who had data from both baseline (pre-treatment) and Part 2 Week 48 (on-treatment) muscle biopsy samples. Data was not planned to be collected and analyzed for untreated group.
Measure: Mean (Standard Deviation); unit: Percent normal dystrophin protein level
Arm/Group | Part 2a: Total Golodirsen Group
Number analyzed (Participants) | 25
Percent normal dystrophin protein level | 0.924 (1.0129)

10. Secondary Outcome: Part 1: Maximum Plasma Concentration (Cmax) of Golodirsen
Description: Maximum Concentration (Cmax) of golodirsen in plasma was evaluated.
Time Frame: Pre-dose, 5 to 10 minutes, 1, 1.5, 2, 4, 6, 8, 12, 16 and 24 hours post-dose at Weeks 1 (for 4 mg/kg arm), 3 (for 10 mg/kg arm), 5 (for 20 mg/kg arm) and 7 (for 30 mg/kg arm)
Population: Pharmacokinetic (PK) set consisted of all randomized participants from Part 1 who received the planned full dose of study drug and for whom there were adequate PK samples from which to estimate PK parameters. Data were not planned to be collected and analyzed for the placebo arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part 1: Golodirsen (4 mg/kg) | Part 1: Golodirsen (10 mg/kg) | Part 1: Golodirsen (20 mg/kg) | Part 1: Golodirsen (30 mg/kg)
Number analyzed (Participants) | 8 | 8 | 8 | 8
nanogram per milliliter (ng/mL) | 7840 (45.7) | 17000 (40.9) | 39700 (71.8) | 53300 (37.9)

11. Secondary Outcome: Part 1: Time to Reach Maximum Plasma Concentration (Tmax) of Golodirsen
Description: Time to reach maximum plasma concentration (Tmax) of golodirsen was evaluated.
Time Frame: as for outcome 10
Population: PK set consisted of all randomized participants from Part 1 who received the planned full dose of study drug and for whom there were adequate PK samples from which to estimate PK parameters. Data were not planned to be collected and analyzed for the placebo arm.
Measure: Median (Full Range); unit: hour
Arm/Group | Part 1: Golodirsen (4 mg/kg) | Part 1: Golodirsen (10 mg/kg) | Part 1: Golodirsen (20 mg/kg) | Part 1: Golodirsen (30 mg/kg)
Number analyzed (Participants) | 8 | 8 | 8 | 8
hour | 1.11 [0.77 to 1.67] | 1.09 [0.12 to 1.62] | 1.12 [0.80 to 1.58] | 1.12 [0.68 to 1.50]

12. Secondary Outcome: Part 1: Area Under the Concentration-Time Curve From Time Zero Extrapolated to the Infinity (AUCinf) of Golodirsen in Plasma
Description: Area under the concentration-time curve from time zero extrapolated to the infinity was evaluated.
Time Frame: as for outcome 10
Population: PK set: all randomized participants from Part 1 who received the planned full dose of study drug and for whom there were adequate PK samples from which to estimate PK parameters. "Overall number of participants analyzed"= number of participants evaluable for this outcome. Data were not planned to be collected and analyzed for the placebo arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Part 1: Golodirsen (4 mg/kg) | Part 1: Golodirsen (10 mg/kg) | Part 1: Golodirsen (20 mg/kg) | Part 1: Golodirsen (30 mg/kg)
Number analyzed (Participants) | 8 | 8 | 6 | 8
hr*ng/mL | 11800 (35.5) | 26400 (42.7) | 62300 (52.6) | 90800 (33.4)

13. Secondary Outcome: Part 1: Apparent Volume of Distribution at Steady State (Vss) of Golodirsen
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution at steady state of golodirsen was evaluated.
Time Frame: as for outcome 10
Population: PK set: all randomized participants from Part 1 who received planned full dose of study drug, for whom there were adequate PK samples from which to estimate PK parameters. "Overall number of participants analyzed"= number of participants evaluable for this outcome. Data were not planned to be collected and analyzed for the placebo arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per kilogram (L/kg)
Arm/Group | Part 1: Golodirsen (4 mg/kg) | Part 1: Golodirsen (10 mg/kg) | Part 1: Golodirsen (20 mg/kg) | Part 1: Golodirsen (30 mg/kg)
Number analyzed (Participants) | 8 | 8 | 6 | 8
Liter per kilogram (L/kg) | 0.670 (38.6) | 0.767 (43.4) | 0.576 (84.5) | 0.668 (32.3)

14. Secondary Outcome: Part 1: Elimination Half-life (T1/2) of Golodirsen
Description: T1/2 is the time measured for the plasma concentration of drug to decrease by one half. T1/2 of golodirsen was evaluated.
Time Frame: as for outcome 10
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Part 1: Golodirsen (4 mg/kg) | Part 1: Golodirsen (10 mg/kg) | Part 1: Golodirsen (20 mg/kg) | Part 1: Golodirsen (30 mg/kg)
Number analyzed (Participants) | 8 | 8 | 6 | 8
hour | 2.36 (0.581) | 3.63 (2.04) | 3.27 (0.897) | 3.42 (0.628)

15. Secondary Outcome: Part 1: Total Clearance (CL) of Golodirsen
Description: Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: as for outcome 10
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Liters per hour per kilogram (L/h/kg)
Arm/Group | Part 1: Golodirsen (4 mg/kg) | Part 1: Golodirsen (10 mg/kg) | Part 1: Golodirsen (20 mg/kg) | Part 1: Golodirsen (30 mg/kg)
Number analyzed (Participants) | 8 | 8 | 6 | 8
Liters per hour per kilogram (L/h/kg) | 0.381 (36.0) | 0.405 (46.2) | 0.338 (52.2) | 0.346 (34.3)

16. Secondary Outcome: Part 1: Mean Residence Time (MRT) of Golodirsen
Description: MRT= AUMCinf/AUCinf, where AUMCinf is the area under the first moment curve from time 0 extrapolated to infinite time, calculated using the linear/log trapezoidal method. Mean residence time of golodirsen was evaluated.
Time Frame: as for outcome 10
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Part 1: Golodirsen (4 mg/kg) | Part 1: Golodirsen (10 mg/kg) | Part 1: Golodirsen (20 mg/kg) | Part 1: Golodirsen (30 mg/kg)
Number analyzed (Participants) | 8 | 8 | 6 | 8
hour | 1.79 (0.325) | 1.92 (0.338) | 1.77 (0.495) | 1.95 (0.312)

17. Secondary Outcome: Part 1: Renal Clearance (CLR) of Golodirsen
Description: Renal clearance was calculated using the partial AUC0-24 from the non-compartmental analysis in plasma and AE0-24. AUC0-24 was defined as area under the plasma concentration-time curve, from time 0 to 24 hours after completion of dosing. AE0-24 was defined as total cumulative amount excreted from 0 to 24 hours. Summarized data of all urine collection intervals are reported.
Time Frame: 0 to 1440 min after initiation of dosing on Day 1
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h/kg
Arm/Group | Part 1: Golodirsen (4 mg/kg) | Part 1: Golodirsen (10 mg/kg) | Part 1: Golodirsen (20 mg/kg) | Part 1: Golodirsen (30 mg/kg)
Number analyzed (Participants) | 8 | 8 | 7 | 8
L/h/kg | 0.345 (31.9) | 0.370 (50.6) | 0.355 (42.1) | 0.374 (26.8)

18. Secondary Outcome: Part 2a: Percent Change From Baseline in Forced Vital Capacity Predicted (FVC%p) at Week144 in Total Golodirsen Group
Description: FVC was the total amount of air exhaled during the forced expiratory volume test that was measured during spirometry and the most important measurement of lung function. This test required participant to breath into a tube connected to a machine that measures the amount of air that can be moved in and out of the lungs after taking an inhaled bronchodilator medicine which was used to dilate participant bronchial (breathing) tubes. Percent of predicted FVC = (observed value)/ (predicted value) * 100%.
Time Frame: Baseline, Week 144
Population: Efficacy set consisted of all randomized participants who had at least 1 post-baseline functional assessment. Here, "overall number of participants analyzed" = number of participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Part 2a: Total Golodirsen Group
Number analyzed (Participants) | 23
Percent change | -8.382 (29.4566)

19. Secondary Outcome: Part 2b: Percent Change From Baseline in Forced Vital Capacity Predicted (FVC%p) at Week144 in Untreated Group (Non-exon 53 Amenable Participants)
Description: FVC was the total amount of air exhaled during the forced expiratory volume test that was measured during spirometry and is the most important measurement of lung function. This test requires participant to breath into a tube connected to a machine that measures the amount of air that can be moved in and out of the lungs after taking an inhaled bronchodilator medicine which was used to dilate participant bronchial (breathing) tubes. Percent of predicted FVC = (observed value)/ (predicted value) * 100%.
Time Frame: Baseline, Week 144
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- Part 2b: Untreated Group (Natural History of Non-exon 53): Untreated participants intended to evaluate the natural history of the disease with DMD and various genetic mutations (not amenable to exon 53 skipping) were included in this group and did not received any treatment. Participants underwent the same study assessments as treated participants in other reporting groups (except for PK sampling and muscle biopsies), but at a reduced schedule through Week 144.Thus, the untreated participants were not considered as control group.
Arm/Group | Part 2b: Untreated Group (Natural History of Non-exon 53)
Number analyzed (Participants) | 5
Percent change | -6.739 (17.5278)

20. Secondary Outcome: Part 2a: Change From Baseline in Dystrophin Intensity Levels Determined by Immunohistochemistry (IHC) at Week 48 in Total Golodirsen Group
Description: Change from baseline in dystrophin Intensity levels (in muscle biopsy samples) was determined by Immunohistochemistry in total golodirsen group.
Time Frame: Baseline, Week 48
Population: Muscle biopsy set included all participants who received at least 1 dose of study drug and who had data from both baseline (pre-treatment) and Part 2 Week 48 (on-treatment) muscle biopsy samples. Data were not planned to be collected and analyzed for the untreated group.
Measure: Mean (Standard Deviation); unit: Percent dystrophin positive fibers
Arm/Group | Part 2a: Total Golodirsen Group
Number analyzed (Participants) | 25
Percent dystrophin positive fibers | 0.023 (0.0243)

21. Secondary Outcome: Part 2a: Percent Change From Baseline in Exon 53 Skipping Determined by Reverse Transcription Polymerase Chain Reaction (PCR) at Week 48 in Total Golodirsen Group
Description: Percent change from baseline in Exon 53 skipping (in muscle biopsy samples) was determined by reverse transcription polymerase chain reaction in total golodirsen group.
Time Frame: Baseline, Week 48
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Part 2a: Total Golodirsen Group
Number analyzed (Participants) | 25
Percent change | 16.363 (10.6223)

22. Secondary Outcome: Part 2a: Percent Change From Baseline in Dystrophin Positive Fibers Determined by Immunohistochemistry (IHC) at Week 48 in Total Golodirsen Group
Description: Percent change from baseline in dystrophin positive fibers (in muscle biopsy samples) were determined by Immunohistochemistry at Week 48 in total golodirsen group.
Time Frame: Baseline, Week 48
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Part 2a: Total Golodirsen Group
Number analyzed (Participants) | 25
Percent change | 12.508 (14.6012)

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to 189 weeks
Arm/Group | Part 1: Placebo | Part 1: Golodirsen (4 mg/kg) | Part 1: Golodirsen (10 mg/kg) | Part 1: Golodirsen (20 mg/kg) | Part 1: Golodirsen (30 mg/kg) | Part 2a: Total Golodirsen Group | Part 2b: Untreated Group (Natural History of Non-exon 53)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/8 | 0/8 | 0/8 | 0/8 | 0/25 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/8 | 0/8 | 0/8 | 0/8 | 4/25 | 2/14
Other Adverse Events (participants affected / at risk) | 4/4 | 5/8 | 5/8 | 3/8 | 6/8 | 25/25 | 10/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Placebo (N=4) | Part 1: Golodirsen (4 mg/kg) (N=8) | Part 1: Golodirsen (10 mg/kg) (N=8) | Part 1: Golodirsen (20 mg/kg) (N=8) | Part 1: Golodirsen (30 mg/kg) (N=8) | Part 2a: Total Golodirsen Group (N=25) | Part 2b: Untreated Group (Natural History of Non-exon 53) (N=14)
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth development disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Placebo (N=4) | Part 1: Golodirsen (4 mg/kg) (N=8) | Part 1: Golodirsen (10 mg/kg) (N=8) | Part 1: Golodirsen (20 mg/kg) (N=8) | Part 1: Golodirsen (30 mg/kg) (N=8) | Part 2a: Total Golodirsen Group (N=25) | Part 2b: Untreated Group (Natural History of Non-exon 53) (N=14)
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 16 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 13 | 4
Gastroenteritis (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 8 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 5 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 3 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 2 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 2
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Scarlet fever (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 15 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 14 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 9 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 9 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Glossitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tooth discolouration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 1 | 1 | 4 | 13 | 1
Abasia (General disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 1
Catheter site bruise (General disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 3 | 0
Infusion site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Catheter site related reaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 9 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 6 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 6 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 6 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 4 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 4 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 4 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 4 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 3 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 3 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3 | 16 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 12 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 6 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 11 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 10 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 9 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 6 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 3 | 11 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 7 | 0
Vitamin D decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Platelet count increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Initial insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Stress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Aggression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 4 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 3 | 0
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The most restrictive relevant agreement provides that the PI can only publish the study results with the approval of Sponsor.

DOCUMENTS (2):
  • Study Protocol (2017-11-08): https://cdn.clinicaltrials.gov/large-docs/06/NCT02310906/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-30): https://cdn.clinicaltrials.gov/large-docs/06/NCT02310906/SAP_001.pdf